CLINICAL TRIAL: NCT02185248
Title: Randomized Controlled Trial of a Wellness Action Plan to Address the Childhood Obesity Epidemic
Brief Title: Wellness Action Plan Trial Addressing Childhood Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roohi Kharofa, MD, MPH (Other)
Responsible Party: Sponsor-Investigator, Roohi Kharofa, MD, MPH, Primary Care Research Fellow, Medical College of Wisconsin
Organization: Medical College of Wisconsin (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 363990-4
Record Dates: First submitted 2014-07-02; First posted 2014-07-09 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Childhood Obesity
Keywords: Pediatric Obesity; Body Mass Index; Weight Perception; Counseling; Health Behavior
MeSH Terms: conditions — Pediatric Obesity; Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): General clinical counseling in regards to child's BMI category and necessary changes to diet and activity regimen.
- Wellness Plan (Experimental): Received a wellness action plan. The plan included a color-coded BMI chart to help parents understand their child's weight category as well as a brief action planning worksheet to help families create personalized plans around healthy diet and activity changes.
  Interventions: Behavioral: Wellness Action Plan

INTERVENTIONS:
Behavioral: Wellness Action Plan — The plan included a color-coded BMI chart to help parents understand their child's weight category as well as a brief action planning worksheet to help families create personalized plans around healthy diet and activity changes.
  Arms: Wellness Plan

SUMMARY:
The objective of this study was to determine the effectiveness of a novel Wellness Action Plan aimed at 1) improving parent recall of diet and activity plans 2) increasing follow-through with plans and 3) aiding parents in identifying their child's weight category.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 2.5 and 14 years, regardless of baseline BMI
* Presented for a well child visit at a pediatric clinic serving primarily Medicaid-insured children in Milwaukee, Wisconsin

Exclusion Criteria:

* Patients in foster care
* Parents and patients who were non-English speaking
* Patients who were being seen by a specialist for weight management.

Ages: 30 Months to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 181 (Actual)
Dates: Start 2013-03; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Diet plan recall directly after visit | On day of primary visit
  Parents are given a questionnaire which asks whether they made a diet plan with their physician for their child during the visit and whether they will attempt to follow-through with the plan made.
Activity plan recall directly after visit | On day of primary visit, directly after seeing physician
  Parents are given a questionnaire which asks whether they made an activity plan with their physician for their child during the visit and whether they will attempt to follow-through with the plan made.

SECONDARY OUTCOMES:
Diet plan recall/follow-through 1 month post visit | 4 weeks after primary visit
  Parents are contacted 4 weeks after their primary visit and given a phone questionnaire which asks whether they made a diet plan with their physician for their child during the last visit and whether they can recall the plan. If parents can recall the plan, they are then asked if they followed-through with the plan (yes, no) and how successful they were with the changes (1-10 scale).
Diet plan recall/follow-through 3 months post visit | 12 weeks after primary visit
  Parents are contacted 12 weeks after their primary visit and given a phone questionnaire which asks whether they made a diet plan with their physician for their child during the last visit and whether they can recall the plan. If parents can recall the plan, they are then asked if they followed-through with the plan (yes, no) and how successful they were with the changes (1-10 scale).
Activity plan recall/follow-through 1 month post visit | 4 weeks after primary visit
  Parents are contacted 4 weeks after their primary visit and given a phone questionnaire which asks whether they made an activity plan with their physician for their child during the last visit and whether they can recall the plan. If parents can recall the plan, they are then asked if they followed-through with the plan (yes, no) and how successful they were with the changes (1-10 scale).
Activity plan recall/follow-through 3 months post visit | 12 weeks after primary visit
  Parents are contacted 12 weeks after their primary visit and given a phone questionnaire which asks whether they made an activity plan with their physician for their child during the last visit and whether they can recall the plan. If parents can recall the plan, they are then asked if they followed-through with the plan (yes, no) and how successful they were with the changes (1-10 scale).
BMI category identification directly after the visit | On day of primary visit
  Parents are given a questionnaire which asks whether their physician told them their child's weight category and asks whether they can identify that category.
BMI category identification 1 month post visit | 4 weeks after primary visit
  Parents are contacted 4 weeks after their primary visit and given a phone questionnaire which asks whether their physician told them their child's weight category and asks whether they can identify that category.
BMI category identification 3 months post visit | 12 weeks after primary visit
  Parents are contacted 12 weeks after their primary visit and given a phone questionnaire which asks whether their physician told them their child's weight category and asks whether they can identify that category.

CONTACTS AND LOCATIONS:
Overall Officials: John R Meurer, MD, MBA, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Downtown Health Center, Milwaukee, Wisconsin, United States

REFERENCES:
- [Derived] Kharofa RY, Copeland KA, Sucharew H, Meurer JR. Randomized controlled trial of a Wellness Action Plan to promote healthy diet and activity in pediatric primary care. Prev Med Rep. 2015 Oct 21;2:899-905. doi: 10.1016/j.pmedr.2015.10.008. eCollection 2015. PMID 26844166